CLINICAL TRIAL: NCT02801084
Title: Examining the Effects of Reduced Environmental Stimulation on Eating Disorders
Brief Title: Effects of Reduced Environmental Stimulation on Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-002-01
Record Dates: First submitted 2016-05-18; First posted 2016-06-15 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2020-10

CONDITIONS: Anorexia Nervosa
Keywords: Reduced; Environmental; Stimulation
MeSH Terms: conditions — Anorexia Nervosa | interventions — Divorce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Float (Experimental): One arm only: restricted environmental stimulation
  Interventions: Behavioral: Reduced environmental stimulation

INTERVENTIONS:
Behavioral: Reduced environmental stimulation — Participants will complete one arm involving four sequential float sessions. Float 1: chair float. Participants will first float in a comfortable chair in the supine position, for up to 90 minutes. The chair is in a room with sound and light attenuation. Orthostatic blood pressure (BP) will be measured before and after each float. Anxiety and body image will be measured afterwards.
  Float 2: open pool float. Participants will float for up to 90 minutes in an open pool (8 foot diameter, no enclosure). Orthostatic BP will be measured before and after each float. Anxiety and body image will be measured afterwards.
  Floats 3 & 4: domed pool float. Participants will float for up to 90 minutes in a domed pool the same size as the open pool, with an enclosure wall and 8 foot tall ceiling. Orthostatic BP will be measured before and after each float. Anxiety and body image will be measured afterwards.
  Each float will occur approximately 1 to 7 days apart.
  Other Names: Floating

SUMMARY:
The study proposed in this protocol aims to document the physiological, subjective, behavioral, and neural effects of reduced environmental stimulation (floating) in patients with current or prior anorexia nervosa The primary aim of this study is to determine the safety of this intervention. Secondary aims including determining whether floating has an impact on symptom reports such as those related to anxiety and eating disorders.

DETAILED DESCRIPTION:
Floating creates an environment with minimal visual, auditory, tactile, proprioceptive, and thermal input to the brain. The float rooms used in this study are both lightproof, and thus completely dark when the entry door is sealed and the lights are turned off, reducing all visual input to the brain. Each float room was constructed with thick soundproof walls, restricting most outside noises from entering the room, thereby reducing auditory input to the brain. A high concentration Epsom salt water solution allows individuals to effortlessly float on their back while remaining completely still, reducing both proprioceptive and tactile input to the brain. The temperature of the water is calibrated to the temperature of the skin (~94° F) and the temperature of the air is calibrated to the temperature of the water, making it difficult to discern the boundary between air and water, thus reducing thermal input to the brain while minimizing the need for thermoregulation of the skin.

While both float pools dramatically reduce external sensory information, it is important to note that participants are in full control over the experience. For example, participants can enter and exit the float pool whenever they choose. Each float pool also contains a blue LED light that can be turned on and off via an air-coupled light switch in the pool. Both float rooms contain a shower for cleaning before and after floating.

In a prior study the investigators have found that healthy participants found the pool condition to be relaxing and stress relieving. The current study aims to determine the safety of floating with a clinical population, specifically individuals with a history of eating disorder who are of normal weight.

ELIGIBILITY:
Inclusion Criteria:

1. Current or prior diagnosis of anorexia nervosa (AN)
2. All AN participants must be weight-restored prior to their participation, defined as having a Body Mass Index (BMI) > 17.5

Exclusion Criteria:

1. Any of the following DSM-V disorders:

   1. Schizophrenia Spectrum and Other Psychotic Disorders
   2. Bipolar and Related Disorders
2. Currently being treated for their psychiatric condition as an inpatient.
3. Active suicidal ideation with intent or plan (as determined by a psychiatrist or clinical psychologist for all participants who report an IDAS-II suicide score > 10).
4. Morbid obesity (BMI > 40) or underweight (BMI < 17.5).
5. Orthostatic hypotension (defined as a drop of ≥20 mm Hg in systolic blood pressure or a drop of ≥10 mm Hg in diastolic blood pressure when measured shortly after transitioning from lying down to standing).
6. Certain drugs or medications consumed within the past week including any psychoactive drugs (e.g., MDMA, LSD, psilocybin, peyote, phencyclidine, ketamine), magnesium supplements (greater than 150mg) or milk of magnesia. Any antihistamine that causes drowsiness (e.g., Benadryl) or any alcohol consumed within the past 12 hours. Caffeine or nicotine consumed within the past 3 hours. For all other medications, participants must be stably medicated prior to participation (defined as having taken the medication for 6 weeks or longer).
7. History of unstable liver or renal insufficiency; glaucoma; diabetes; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance.
8. Pregnancy as detected by a urine test.
9. Failure to adhere to "Pre-float checklist".
10. Non-correctable vision or hearing problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Orthostatic blood pressure | Immediately before and after each float session for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Defined as a drop of ≥20 mm Hg in systolic blood pressure or a drop of ≥10 mm Hg in diastolic blood pressure when measured shortly after transitioning from lying down to standing.

SECONDARY OUTCOMES:
Self-ratings of changes in emotional experience | Immediately before and after each float session for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Measured via self-report measure (Positive and Negative Affect Schedule X)
Self-ratings of changes in physical experience | Immediately before and after each float session for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Interoceptive and exteroceptive sensations, measured via visual analogue scale (e.g., 0 to 100)
Body image | Obtained at baseline and immediately after each float session for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Measured via Photographic Figure Rating Scale, Body Appreciation Scale, Body Image States Scale, Body Shape Questionnaire, visual analogue scale (e.g., 0 to 10).
EEG changes during the float experience | During the first, second, and fourth float for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  May be measured during the first, second, and fourth float.
Heart rate variability during the float experience | Obtained at baseline and after the first, second, and fourth float for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Measured during the first, second, and fourth float.
Eating disorder severity | Obtained during the first visit
  Measured via the Eating Disorder Examination Questionnaire
Trauma exposure | Obtained during the first visit
  Measured via the Childhood Trauma Questionnaire
Self-ratings of changes in anxiety | Obtained at baseline and immediately before and after each float session for 4 float sessions, spaced weekly to monthly for up to 16 weeks study duration
  Measured via self-report measure (Spielberger State-Trait Anxiety Index)
Self-ratings of anxiety sensitivity | Obtained during the first visit
  Measured via the Anxiety Sensitivity Index

CONTACTS AND LOCATIONS:
Overall Officials: Sahib S Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Khalsa SS, Moseman SE, Yeh HW, Upshaw V, Persac B, Breese E, Lapidus RC, Chappelle S, Paulus MP, Feinstein JS. Reduced Environmental Stimulation in Anorexia Nervosa: An Early-Phase Clinical Trial. Front Psychol. 2020 Oct 6;11:567499. doi: 10.3389/fpsyg.2020.567499. eCollection 2020. PMID 33123048
- See also: DOI for publication summarizing study results. — https://doi.org/10.3389/fpsyg.2020.567499